CLINICAL TRIAL: NCT01710761
Title: Effects of Neo40(TM) With Caffeine on Cycling Time Trial Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Neogenis Laboratories (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012-05-0033
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: nitric oxide; cycling performance; lactate; VO2
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrate supplement with caffeine (Active Comparator)
  Interventions: Dietary Supplement: Nitrate supplement with caffeine
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Same form factor and flavor as test lozenge but contains no active ingredients
  Arms: Placebo
Dietary Supplement: Nitrate supplement with caffeine — Lozenge consisting of beetroot and 75 mg caffeine
  Arms: Nitrate supplement with caffeine

SUMMARY:
Acute supplementation of Neo40(TM), a nitrate lozenge, will improve cycling performance

ELIGIBILITY:
Inclusion Criteria:

* Regular commuter cyclist or spin class participant
* Male (VO2max < 50) or Female (VO2max < 45)
* Healthy
* Blood pressure below 140/90
* Non-smoker

Exclusion Criteria:

* Does not cycle 2-3 times/week
* Regular consumption of performance-enhancing substances
* Type I or Type II diabetes
* Renal, hepatic or cardiac disease
* Current infectious disease

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-02 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Improved Time Trial Performance | After 20 min steady-state cycling
  Participants will cycle 20 min at increasing intensity: 8 min at 55% VO2max, 6 min at 65% VO2max, 6 min at 75% VO2max. The 20 km time trial consists of rolling hills.

SECONDARY OUTCOMES:
Improved work efficiency | During 20 min steady-state cycling
  Expired gases will be collected and compared to expected VO2. Blood will be collected prior to treatment, prior to exercise and during each cycling intensity to analyze lactate accumulation.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Kammer-Kerwick, MSE, MA, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States